CLINICAL TRIAL: NCT01060475
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Exploratory Pharmacodynamics of LIM-0705 Given With or Without Tacrolimus in Healthy Male Subjects
Brief Title: Safety and Tolerability of LIM-0705 in Healthy Male Subjects
Acronym: LIM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Limerick BioPharma (Industry)
Responsible Party: Wendye Rae Robbins, MD, Limerick BioPharma
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIM-0705-CL-002
Record Dates: First submitted 2010-01-29; First posted 2010-02-02 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Transplant
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Experimental): Low dose LIM-0705 and tacrolimus.
  Interventions: Drug: LIM-0705 and tacrolimus
- B (Experimental): High dose LIM-0705 and tacrolimus.
  Interventions: Drug: LIM-0705 and tacrolimus
- C (Experimental): Placebo LIM-0705 and tacrolimus.
  Interventions: Drug: Placebo LIM-0705 and tacrolimus
- D (Experimental): High dose LIM-0705 and placebo tacrolimus.
  Interventions: Drug: Drug LIM-0705 and placebo tacrolimus

INTERVENTIONS:
Drug: LIM-0705 and tacrolimus — Oral solution, LIM-0705 500 mg BID for 14 days plus tacrolimus BID for first 8 days.
  Arms: A
Drug: LIM-0705 and tacrolimus — Oral solution, LIM-0705 750 mg BID for 14 days plus tacrolimus BID for the first 8 days.
  Arms: B
Drug: Placebo LIM-0705 and tacrolimus — Placebo oral solution BID for 14 days plus tacrolimus BID for the first 8 days.
  Arms: C
Drug: Drug LIM-0705 and placebo tacrolimus — Oral solution, LIM-0705 750 mg BID for 14 days plus placebo capsule BID for the first 8 days.
  Arms: D

SUMMARY:
LIM-0705 dosed separately and in combination with tacrolimus will be safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Male age 18-50
* Patient in good health as deemed by pre-study exam and history
* BMI 20-30 kg/sq. meter
* Absence of tremors
* Must be willing to remain in confinement for 17 days/16 nights
* Systolic BP 90-140 mmHg, diastolic BP 50-90 mmHg, resting HR 45-90 bpm
* Subject must be non-smoker or willing to abstain from smoking day -4 through day 30.
* Subject must abstain from alcohol, grapefruit,and caffeine-containing beverages starting Day -2 through Day 30.
* Subjects must use double-barrier contraception through course of study + 90 days following study

Exclusion Criteria:

* Allergy to red wine or onions
* Strict vegetarians
* Use of any non-study medication
* Use of chemotherapy within 5 years prior to Screening visit
* Use of any dietary aids
* Difficultly swallowing oral medications
* cognitive or psychiatric disorders

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of LIM-0705 with and without co-administered drug (tacrolimus). | 14 days

SECONDARY OUTCOMES:
Pharmacokinetics of LIM-0705 with and without combination of co-administered drug (tacrolimus). | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Albert Frauman, MD, Study Director — Nucleus Network
Locations (2):
- Australia (2):
  - Nucleus Network CCS-Austin, Heidelberg, Victoria
  - Nucleus Network CCS-AMREP, Prahran, Victoria